CLINICAL TRIAL: NCT02001896
Title: A Randomized, Open-label Phase III Study of First-line Treatment With Erlotinib Intercalated With Gemcitabine/ Cisplatin or Carboplatin Therapy Versus Erlotinib in Stage IIIB/IV NSCLC Patients With EGFR Mutation
Brief Title: Erlotinib Intercalated With Chemotherapy Versus Erlotinib as First Line Treatment in Stage IIIB/IV NSCLC Patients With EGFR Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, li shan, chief physician, Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTHLC001
Record Dates: First submitted 2013-11-21; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; EGFR-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Carboplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- erlotinib combine with chemotherapy (Experimental): Drug: gemcitabine 1000mg/m2 iv on days 1 of each 4 week cycle for 6 cycles Drug: Platinum chemotherapy (cisplatin or carboplatin) cisplatin --75mg/m2 oon day 1 of each 4 week cycle for 6 cycles or carboplatin--5xAUC on day 1 of each 4 week cycle for 6 cycles Drug: Erlotinib[Tarceva] po on days 15-28 of each 4 week cycle until disease progression
  Interventions: Drug: gemcitabine; cisplatin or carboplatin; erlotinib
- erlotinib along (Active Comparator): Drug: erlotinib [Tarceva] 150mg/day po until disease progression
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: gemcitabine; cisplatin or carboplatin; erlotinib
  Other Names: tarceva
  Arms: erlotinib combine with chemotherapy
Drug: erlotinib
  Other Names: tarceva
  Arms: erlotinib along

SUMMARY:
This 2 arm study will compare the efficacy and safety of treatment with erlotinib intercalated with platinum-based therapy or erlotinib along, as first line treatment in Stage IIIB/IV Non-Small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor (EGFR) Mutation. Patients will be randomized to receive gemcitabine (1000mg/m2 iv) on days 1 , and cisplatin (75mg/m2) or carboplatin (5xAUC)on day 1, followed by erlotinib 150mg/day from day 15 to day 28 of each 4 week cycle for a total of 6 cycles,then followed by erlotinib monotherapy, or erlotinib 150mg/day .The anticipated time on study treatment is until disease progression, and the target sample size is 60 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;advanced (stage IIIB/IV)non-small cell lung cancer;measurable disease;ECOG Performance Status 0-2.

Exclusion Criteria:

* prior exposure to agents directed at the HER axis;prior chemotherapy or systemic anti-tumor therapy after advanced disease;unstable systemic disease; any other malignancy within last 5 years, except cured basal cell cancer of skin or cured cancer in situ of cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 24 mont

CONTACTS AND LOCATIONS:
Locations (1):
- Xinjiang medical university, Ürümqi, Xinjiang, China